CLINICAL TRIAL: NCT01198028
Title: Phase II Study of Erlotinib, An Epidermal Growth Factor Receptor (EGFR) Tyrosine Kinase Inhibitor, in the Treatment of Recurrent or Metastatic Squamous Cell Carcinoma of the Skin
Brief Title: Erlotinib in Treating Patients With Recurrent or Metastatic Skin Squamous Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0888; NCI-2018-01834 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2009-0888 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2010-09-08; First posted 2010-09-09 (Estimated); Results first posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Metastatic Skin Squamous Cell Carcinoma; Recurrent Skin Squamous Cell Carcinoma
MeSH Terms: interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (erlotinib) (Experimental): Participants receive erlotinib PO QD in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib — Given PO

SUMMARY:
This phase II trial studies how well erlotinib works in treating participants with skin squamous cell carcinoma that has spread to other places in the body or has come back. Drugs used in chemotherapy, such as erlotinib, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the overall response rate with erlotinib in patients with locoregionally recurrent or metastatic squamous cell carcinoma of the skin (CSCC) that is not amenable to curative treatment.

SECONDARY OBJECTIVES:

I. To determine duration of response and duration of stable disease. II. To determine progression-free and overall survival. III. To determine safety and tolerability of erlotinib.

EXPLORATORY OBJECTIVES:

I. To correlate baseline expression of estimated glomerular filtration rate (EGFR), expression of markers of EGFR activation (such as phosphorylated [p] EGFR and pAKT) and related cell-signaling pathways, and EGFR mutation status with response to erlotinib therapy.

II. To determine the effects of erlotinib on relevant biomarkers of the EGFR pathway in tumor tissue and in normal skin, and to correlate with response to therapy.

III. To determine if there is a correlation between the development of erlotinib-induced skin rash and response to therapy.

OUTLINE:

Participants receive erlotinib orally (PO) once daily (QD) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically or cytologically confirmed cutaneous squamous cell carcinoma (CSCC) that is not amenable to curative therapy. If the biopsy was collected outside of MD Anderson Cancer Center (MDACC), the MDACC Pathology Department must assess and confirm the squamous cell carcinoma (SCC) diagnosis.
* Have measurable disease.
* Have Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Must have ability to understand and the willingness to sign a written Informed Consent Document (ICD). In the event that non-English speaking participants are eligible for this study, a short form (if applicable) or an ICD in their language will be utilized and completed in accordance with the MDACC "Policy For Consenting Non-English Speaking Participants.
* Leukocytes >= 3,000/mm^3.
* Absolute neutrophil count >= 1,500/mm^3.
* Platelets >= 75,000/mm^3.
* Hemoglobin >= 8g/dL.
* Total bilirubin =< 2 x institutional upper limit of normal (ULN).
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 x ULN if alkaline phosphatase is normal, or alkaline phosphatase =< 4 x ULN if transaminases are normal.
* Creatinine =< 2.0 x ULN or creatinine clearance >= 60 mL/min/1.73 m^2.
* Prior radiotherapy is allowed if: (a) there is measurable disease outside the radiation field OR (b) radiotherapy was completed more than 4 weeks ago and there is clearly recurrent and growing disease within the radiation field.
* Must be able to take intact tablets by mouth, or be able to take tablets dissolved in water by mouth or by a percutaneous gastrostomy tube.
* Patients - both males and females - with reproductive potential (includes women who are menopausal for less than 1 year and not surgically sterilized) must practice effective contraceptive measures such as barrier methods, condom or diaphragm with spermicide, or abstinence throughout the study. Birth control should continue for 4 weeks after discontinuation of erlotinib therapy. Women of childbearing potential must provide a negative pregnancy test (serum beta human chorionic gonadotropin [HCG]) within 72 hours prior to first receiving protocol therapy.
* Organ transplant patients are eligible as long as they do not have active signs of rejection and have adequate bone marrow function.

Exclusion Criteria:

* Women who are pregnant, breastfeeding, and women and men not practicing effective birth control. Erlotinib is a signal transduction inhibitor agent with the potential for teratogenic or abortifacient effects. There is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with erlotinib. Breastfeeding should be discontinued if the mother is treated with erlotinib.
* Prior estimated glomerular filtration rate (EGFR) inhibitor therapy is not allowed (including, but not limited to, erlotinib, gefitinib, cetuximab, panitumumab, vandetanib).
* Patients who are receiving any other anticancer or investigational agents at time of study enrollment. Patients may have received one other systemic therapy or investigational agent in the past, but a washout time period of at least 4 weeks and recovery of any treatment-related toxicities to < Common Terminology Criteria for Adverse Events version 4 (CTCAEv4) grade 2 is required.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to erlotinib.
* Patients with a history of an invasive malignancy (other than the one treated in this study) or lymphoproliferative disorder within the past 3 years. Patients with a history of adequately treated non-melanoma skin cancer, ductal carcinoma in situ of the breast, or carcinoma in situ of the cervix are allowed.
* Patients with incomplete healing from previous surgery.
* Patients with pulmonary fibrosis (other than in a radiated field) or active interstitial lung disease.
* Patients with active gastrointestinal disease or a disorder that alters gastrointestinal motility or absorption, including lack of integrity of the gastrointestinal tract (for example, a significant surgical resection of the stomach or small bowel, inflammatory bowel disease or uncontrolled chronic diarrhea.
* Patients with skin rash CTCAEv4 grade 2.
* In the opinion of the investigator, patients with any condition that is unstable or could jeopardize the safety of the patient or could limit compliance with the study's requirements. These include, but are not limited to, ongoing or active infection requiring parenteral antibiotics at time of study registration, psychiatric illness that would limit compliance with study requirements or symptomatic congestive heart failure (New York Heart Association [NYHA] class II or greater), unstable angina pectoris or cardiac arrhythmia requiring maintenance medication.
* Patient is unwilling or unable to discontinue prohibited concomitant therapies, (i.e St. John's wort, grapefruit juice, histamine type 2 receptor [H2] blockers/proton pump inhibitors, strong CYP3A4 inhibitors and inducers).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-03-10 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Glisson, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Gold KA, Kies MS, William WN Jr, Johnson FM, Lee JJ, Glisson BS. Erlotinib in the treatment of recurrent or metastatic cutaneous squamous cell carcinoma: A single-arm phase 2 clinical trial. Cancer. 2018 May 15;124(10):2169-2173. doi: 10.1002/cncr.31346. Epub 2018 Mar 26. PMID 29579331
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in head and neck clinic and from referrals from outside clinics between April 2011 and June 2014 at MD Anderson Cancer Center.
Pre-assignment Details: A total of 42 participants enrolled,39 participants started 1 withdrew, 1 came off study the same day consented and 1 participant was ineligible.
Groups:
- Erlotinib: 150 mg once daily by mouth.
Period: Overall Study
Arm/Group | Erlotinib
Started | 39
Completed | 29
Not Completed | 10
Not completed — Adverse Event | 5
Not completed — Death | 3
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Erlotinib
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 37
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall response rate defined as the percentage of patients who achieve an overall response of complete response or partial response in the total number of evaluable patients, assessed by Response Evaluation Criteria in Solid Tumors 1.1A Bayesian design based on predictive probability will be implemented.
Time Frame: up to 6 years
Measure: Count of Participants; unit: Participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 29
Participants | 3

2. Secondary Outcome: Duration of Response
Description: The time from initial response during therapy to progression of disease evaluated using Kaplan-Meier estimation techniques.
Time Frame: up to 6 years
Measure: Median (Full Range); unit: months
Arm/Group | Erlotinib
Number analyzed (Participants) | 29
months | 5.3 [4.6 to 13.2]

3. Secondary Outcome: Duration of Stable Disease
Description: The date of stable disease to the date of loss of stable disease or last follow-up.
Time Frame: up to 6 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib
Number analyzed (Participants) | 39
months | 7.2 [1.6 to 41.4]

4. Secondary Outcome: Progression-free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: up to 6 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib
Number analyzed (Participants) | 39
months | 4.7 [3.5 to 6.2]

5. Secondary Outcome: Overall Survival
Description: Time from date of treatment start until date of death due to any cause or last Follow-up.
Time Frame: up to 6 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib
Number analyzed (Participants) | 39
months | 13 [8.4 to 20.5]

6. Secondary Outcome: Number of Participants With Safety and Tolerability of Erlotinib
Description: Frequency of adverse events according to the NCI Common Toxicity Criteria for Adverse Effects (CTCAE) v4.0. Standard reporting guidelines followed for adverse events.
Time Frame: Baseline start of treatment, up to 30 days after treatment or to death, up to 6 years
Measure: Count of Participants; unit: Participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 39
Participants
  Dry eyes | 4
  Watery eyes | 10
  Constipation | 5
  Nausea/Vomitting | 10
  Oral Mucositis | 8
  Fatigue | 14
  Acneiform rash | 22

ADVERSE EVENTS:
Time Frame: up to 6 years
Arm/Group | Erlotinib
All-Cause Mortality (participants affected / at risk) | 7/39
Serious Adverse Events (participants affected / at risk) | 7/39
Other Adverse Events (participants affected / at risk) | 22/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=39)
Alanine aminotransferase increased (Investigations) | 1
Lung Infection (Infections and infestations) | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Anemia (grade 3) (Blood and lymphatic system disorders) | 1
Nausea (grade 3) (Gastrointestinal disorders) | 1
Diarrhea (grade 3) (Gastrointestinal disorders) | 1
Vomitting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=39)
Acneiform rash (Skin and subcutaneous tissue disorders) | 22
Fatigue (General disorders) | 14
Dry eyes (Eye disorders) | 4
Oral Mucositis (Gastrointestinal disorders) | 8
Nausea/Vomiting (Gastrointestinal disorders) | 10
Constipation (Gastrointestinal disorders) | 5
Watery eyes (Eye disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-03): https://cdn.clinicaltrials.gov/large-docs/28/NCT01198028/Prot_SAP_000.pdf